CLINICAL TRIAL: NCT01982201
Title: A Phase 1, Randomized, Open-Label, Drug-Drug Interaction Study to Evaluate the Potential Pharmacokinetic and Pharmacodynamic Interaction Between Lesinurad and Calcium Carbonate and Aluminum/Magnesium Hydroxide-Containing Antacids in Healthy Adult Male Subjects
Brief Title: Antacid Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA594-130
Record Dates: First submitted 2013-11-08; First posted 2013-11-13 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — lesinurad; Calcium Carbonate; aluminum hydroxide, magnesium hydroxide, simethicone drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lesinurad and Tums (Experimental): Day 1: 240 mL water or 240 mL water and Tums Day 2: Lesinurad 400 mg or Lesinurad 400 mg and Tums; Day 6: 240 mL water and Tums or 240 mL water; Day 7: Lesinurad 400 mg and Tums or Lesinurad 400 mg
  Interventions: Drug: Lesinurad 400 mg; Drug: Tums 500 mg and 750 mg
- Lesinurad and MINTOX (Experimental): Day 1: 240 mL water or 240 mL water and MINTOX ; Day 2: Lesinurad 400 mg or Lesinurad 400 mg and MINTOX; Day 6: 240 mL water and MINTOX or 240 mL water; Day 7: Lesinurad 400 mg and MINTOX or Lesinurad 400 mg
  Interventions: Drug: Lesinurad 400 mg; Drug: MINTOX 10 mL

INTERVENTIONS:
Drug: Lesinurad 400 mg
Drug: Tums 500 mg and 750 mg
  Arms: Lesinurad and Tums
Drug: MINTOX 10 mL
  Arms: Lesinurad and MINTOX

SUMMARY:
This study will assess the potential effects of calcium carbonate and aluminum/magnesium hydroxide-containing antacids on the pharmacokinetics (PK) and pharmacodynamics (PD) of lesinurad in healthy, adult male subjects.

DETAILED DESCRIPTION:
In this study, lesinurad and antacid will be administered in the fed state, antacid doses will be attenuated to reflect the more commonly used doses, baseline PD assessments will be performed both in presence and absence of antacid treatment, and the sequence of treatments (lesinurad +/- antacid) will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body weight ≥ 50 kg (110 lbs) and body mass index ≥ 18 and ≤ 30 kg/m2.
* Subject is free of any clinically significant disease or medical condition, per the Investigator's judgment

Exclusion Criteria:

* Subject has a history or suspicion of kidney stones.
* Subject has undergone major surgery within 3 months prior to Screening.
* Subject donated blood or experienced significant blood loss (>450 mL) within 12 weeks prior to Screening or gave a plasma donation within 4 weeks prior to Screening.
* Subject has inadequate venous access or unsuitable veins for repeated venipuncture.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
PK profile of lesinurad from plasma and urine | Day 2 and Day 7
  Plasma in terms of maximum observed concentration (Cmax), time of occurrence of maximum observed concentration (Tmax), area under the concentration-time curve (AUC), apparent terminal half-life (t½), renal clearance (CLR), and adverse event (Ae).
PD profile of Lesinurad from serum and urine | Day 2 and Day 7
  Serum PD in terms of serum urate concentration, urine uric acid excretion amount, renal clearance of uric acid, and fractional excretion of uric acid.

SECONDARY OUTCOMES:
Incidence of Adverse Events and Changes in Laboratory, Electrocardiogram, and Vital Signs Parameters | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Kalamazoo, Michigan, United States